CLINICAL TRIAL: NCT05923580
Title: Group-based Cardiac Telerehabilitation and Its Effectiveness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Oulu University Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University of Eastern Finland
Record Dates: First submitted 2023-06-05; First posted 2023-06-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Cardiac telerehabilitation; Quality of life; Adherence to treatment; Lifestyle change
MeSH Terms: conditions — Coronary Artery Disease; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Participants' quality of life (measured with the 15D quality of life instrument), lifestyle changes, and adherence to treatment will be measured using quantitative methods with a quasi-experimental research design and interrupted time- series design. The power analysis for the study will be conducted using Finnish population norms for the 15D instrument. The sample size will be 198 cardiac rehabilitation participants (N=198), with 99 participants in the intervention group (N=99) and 99 participants in the control group (N=99). With this sample size, a power of over 80% (p=0.05) will be achieved to detect a difference of 0.12 (0.95 vs. 0.83, SD=0.3) in quality of life between the groups.
Masking Description: All the participants are being treated in a healthcare unit that uses digital care pathways for coronary patients. Patients can choose the usual care or group-based cardiac telerehabilitation as follow-up care. All the patients are invited to the study after the chosen follow-up care (telerehabilitation or usual care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goup-based cardiac telerehabilitation (Experimental): Group-based cardiac telerehabilitation promotes information, skills, and support for the management of coronary artery disease in coronary patients. The rehabilitation model includes independent familiarization with information content, assignments, and group meetings, as well as the opportunity for a chat and peer support. The intervention is a health professional- lead, and registered rehabilitation model with a start and end.
  Interventions: Behavioral: Group- based cardiac telerehabilitation
- Usual care for cardiac patients (No Intervention): The coronary patient is in primary care under the supervision of a nurse and a doctor.

INTERVENTIONS:
Behavioral: Group- based cardiac telerehabilitation — Group-based cardiac telerehabilitation promotes information, skills, and support for the management of coronary artery disease in coronary patients. The rehabilitation model includes independent familiarization with information content, assignments, and group meetings, as well as the opportunity for a chat and peer support. The intervention is a health professional- lead, and registered rehabilitation model with a start and end.
  Other Names: Tulppa- telerehabilitation
  Arms: Goup-based cardiac telerehabilitation

SUMMARY:
Cardiovascular diseases (CVD) and coronary artery diseases (CAD) are the most common cause of death worldwide. After an acute cardiac event, prevention of new cardiac events is essential and reduces suffering. Group-based cardiac telerehabilitation (CTR) refers to the use of information and communication technologies for rehabilitation purposes in promoting CAD patients´ health.

DETAILED DESCRIPTION:
This study aims to assess the group-based cardiac telerehabilitation model and its effectiveness. The data is collected from two University hospitals in Finland. Patients with coronary heart disease two months after percutaneous coronary intervention (N=198) are invited to the study. All the participants are being treated in a healthcare unit that uses digital care pathways for coronary patients. Patients can choose the usual care or group-based cardiac telerehabilitation as follow-up care. All the patients are invited to the study after the chosen follow-up care (telerehabilitation or usual care). Patients will be allocated into two groups: The telerehabilitation group is the intervention group and the usual care group is the control group. Quality of life, adherence to treatment, and lifestyle changes are measured at the baseline and 3, 6, and 12 after the intervention baseline.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have patients with coronary heart disease two months after percutaneous coronary intervention.
* Participants must have ≥18 years of age, and ≤100 years of age
* Participants are being treated in a healthcare unit that uses digital care pathways for coronary patients.

Exclusion Criteria:

* Participants must not have coronary artery disease diagnosed.
* Participants have been in other operations than percutaneous coronary intervention.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men, women, other gender, do not want to tell
Enrollment: 198 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in The health-related quality of life at 12 Months | Baseline and 12 Months
  15D The health-related quality of life (HRQoL) instrument is a generic, comprehensive (15-dimensional), self-administered instrument for adults (age 16+ years). It combines the advantages of a profile and a preference-based, single index measure. A set of utility or preference weights is used to generate the 15D score (single index number) on a 0-1 scale, representing the overall HRQoL (0 = being dead, 0.0162 = being unconscious or comatose, 1 = no problems on any dimension = 'full' HRQOL). Change = (Month 12 score- Baseline score).
Change from Baseline in The Adherence to Treatment at 12 Months | Baseline and 12 Months
  Adherence to Treatment is a self-assessment instrument designed to describe adherence to treatment of long-term conditions. The questionnaire contains 38 items of adherence to treatment, which are rated on a 5-point Likert scale ('definitely disagree' to 'definitely agree').
Change from Baseline in The Adherence to Medication at 12 Months | Baseline and 12 Months
  Adherence to Medication- instrument is a generic, self-administered instrument. The questionnaire contains items of adherence to medication, which are rated on a 5-point Likert scale ('definitely disagree' to 'definitely agree').
Change from Baseline in Health and Well- being at 12 Months | Baseline and 12 Months
  Health and well-being - the instrument is a generic, self-administered instrument. The questionnaire contains items on the factors influencing health and well-being (smoking, use of alcohol, eating habits, physical activity, sleep), which are rated on a 5-point Likert scale ('definitely disagree' to 'definitely agree').

CONTACTS AND LOCATIONS:
Locations (1):
- Renuka Julia Jacobsson, Tuusula, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No